CLINICAL TRIAL: NCT01452854
Title: Ovarian Aging in Women Newly Diagnosed With Low Grade Glioma Treated With Temozolomide (Temodar®)
Brief Title: Ovarian Aging in Low Grade Glioma (LGG) Treated With Temozolomide
Acronym: OVA-LGG
Status: Terminated | Type: Observational
Why Stopped: Low recruitment, sponsor withdrew funding.
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: UCSF 10-03288
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Low Grade Glioma
Keywords: LGG; Temozolomide; Temodar; Ovarian Aging; Infertility; Chemotherapy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer: The study cohort will include adult women of childbearing potential with a diagnosis of low grade glioma (WHO grade II) who are being treated with low doses of Temozolomide (Temodar).

SUMMARY:
The purpose of this study is to look at how a chemotherapy treatment (Temozolomide, also called Temodar) affects the process of ovarian aging which is measured by a decline in ovarian follicle count, in patients with Low Grade Glioma (LGG). It is important to know if different patient factors and Temozolomide influence the rate of ovarian aging in women with LGG who have good long-term survival rates. This will allow better counseling about the effects of this particular chemotherapy agent on fertility in women.

DETAILED DESCRIPTION:
Understanding how Temozolomide influences ovarian aging would be important information for physicians to predict the possibility of infertility (the inability to become pregnant) following recovery from Temozolomide treatment. Physicians would like to provide better individualized recommendations for cancer patients regarding timing of planned treatment and future pregnancy.

We will do this by comparing data from the women being treated for Low Grade Glioma with Temozolomide to a similar group of women who have been unaffected by cancer or cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women ages 18-44 newly diagnosed with LGG
* Patients fulfill the inclusion criteria for UCSF Protocol Number: CC #99102 " A Phase II Study of Temozolomide (TEMODAR) in the Treatment of Adult Patients with Supratentorial Low Grade Glioma"
* Patients with histologically proven supratentorial low grade glioma.
* Patients may or may not have had a surgical resection.
* Patients must be expected to live the length of study
* Patients must be able to provide informed consent according to institutional guidelines.

Exclusion Criteria:

* Prior ovarian resection, unilateral or bilateral oophorectomy, hysterectomy or radiation to pelvic region.
* Pregnancy or breast feeding.
* Diagnosis of another malignancy, unless the patient was diagnosed at least 2 years earlier and has been disease-free for at least 6 months following the completion of curative intent therapy with the following exceptions: Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study cohort will include adult women of childbearing potential with a diagnosis of low grade glioma (WHO grade II) who are being treated with temozolomide (Temodar).
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — UCSF Center for Reproductive Health and Fertility Preservation; Michael Prados, MD, Study Director — UCSF Department of Neurological Surgery and Helen Diller Comprehensive Cancer Center
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Low recruitment necessitated the closing of the study. No results available.
Period: Overall Study
Arm/Group | Cancer
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Low recruitment necessitated the closing of the study. No results available.
Arm/Group | Cancer
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Ovarian Aging (AFC and Hormones)
Description: Transvaginal Ultrasound will be use to measure Antral Follicle Counts (AFC) and blood will be drawn to measure hormones (FSH, LH, estradiol, estrone, AMH, SHBG, testosterone, and inhibin B).
Time Frame: Every 3 months for 1 year
Population: Data collection was terminated and analyses were not performed due to low enrollment
Arm/Group | Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: This is a non-treatment study so there was no reporting of AEs. Adverse events due to temozolomide treatment, if any, were handled as per institutional guidelines and the Cancer Center protocols.
Groups:
- Cancer: The study cohort will include adult women of childbearing potential with a diagnosis of low grade glioma (WHO grade II) who are being treated with low doses of Temozolomide (Temodar).
  Low recruitment necessitated the closing of the study. No results available.
Arm/Group | Cancer
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No